CLINICAL TRIAL: NCT00003861
Title: Molecular Genetic Features of Acute Leukemia
Brief Title: Diagnostic Study of Patients With Acute Lymphoblastic Leukemia or Acute Promyelocytic Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9862; U10CA076001 (NIH); CALGB-9862; CDR0000067025 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia; Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, Blood

GROUPS / COHORTS (1):
- Ancillary-Correlative (molecular genetic features): Previously collected blood and tissue samples are analyzed via RT-PCR and flow cytometry.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
This research trial studies molecular genetic features in blood and tissue samples from patients with newly diagnosed acute lymphoblastic leukemia or acute promyelocytic leukemia. Studying samples of blood and tissue from patients with acute lymphoblastic leukemia or acute promyelocytic leukemia in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
Objectives:

1. To perform quantitative PCR using known leukemia specific markers in diagnostic bone marrow specimens of patients with newly diagnosed APL and ALL and to correlative pre-treatment copy number with other biologic and molecular features, clinical response, and treatment outcome.
2. To evaluate the expression of novel genes or microRNAs implicated in disease pathogenesis and treatment response in pretreatment blood and bone marrow specimens of patients with APL and ALL and to correlate expression level with other biological features and treatment outcome.
3. To evaluate the clinical significance of sequential quantitative MRD measurements using real-time quantitative PCR and/or flow cytometry during and following treatment of ALL and APL and correlate these findings with efficacy of novel treatment approaches and with other biological and clinical prognostic features.
4. To compare measurement of MRD in blood with bone marrow specimens in sequential remission specimens of patients receiving treatment on ALL and APL treatment trials.

ELIGIBILITY:
* Patients with a diagnosis of acute lymphoblastic leukemia (ALL) entered onto CALGB treatment trials for previously untreated ALL must be enrolled on CALGB 9862. Entry on CALGB 8461 is strongly encouraged.
* Patients with a diagnosis of acute promyelocytic leukemia (APL) enrolled on SWOG S0521 or S0535 must be enrolled on CALGB 9862.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled on CALGB-19802, any CALGB treatment trial, SWOG-S0521, or SWOG-S0535
Sampling Method: Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 1999-04; Primary Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | At baseline
Overall survival | At baseline
Association of novel genes or micorRNAs with other biomarkers | At baseline

SECONDARY OUTCOMES:
Clinical significance of minimal residual disease (MRD) as defined by BCR-ABL | At baseline
Clinical significance of MRD as defined by W T-1 | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Study Chair — University of Chicago
Locations (51):
- United States (51):
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia